CLINICAL TRIAL: NCT01478854
Title: A Prospective Trial of Neural Progenitor Cell Sparing Radiation Therapy Plus Temozolomide for Newly Diagnosed Glioblastoma Multiforme
Brief Title: Neural Progenitor Cell Sparing Radiation Therapy Plus Temozolomide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J10100; NA_00042009 (Other: JHM IRB)
Record Dates: First submitted 2011-11-03; First posted 2011-11-23 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Radiation; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neural Progenitor Cell Sparing Radiation with Temozolomide (Experimental): All subjects are treated with neural progenitor cell sparing radiation to 60 Gy in 2 Gy per day, 30 fractions Concurrent and adjuvant temozolomide chemotherapy
  Interventions: Radiation: Radiation; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Radiation — Patients will be treated to a total dose of 60 Gy with a once daily fractionation schedule of 2 Gy per fraction, administered five days per week. All patients will undergo CT simulation with intravenous contrast. In addition they will undergo MRI simulation with both T1 with gadolinium as well as FLAIR sequences. They will be treated in a supine position using an aquaplast mask system for immobilization. CT image data will be reconstructed in approximately 3 mm slice thickness and manually coregistered with T1 post-gadolinium and FLAIR sequence MRI.
Drug: Chemotherapy — Temozolomide

SUMMARY:
The long term goal of this research is to establish whether NPC sparing RT techniques improve neurocognitive outcomes compared to conventional RT for brain tumors. If the proposed study demonstrates that NPC sparing RT is not associated with increased LR in the spared regions of the brain compared to conventional RT, it will ideally serve as the foundation for a future multi-institutional randomized controlled trial comparing neurocognitive outcomes in patients treated with NPC-sparing RT versus conventional radiation therapy.

DETAILED DESCRIPTION:
Radiation therapy (RT) is an integral component of the management of brain tumors, but cognitive deficits following cranial irradiation are well documented. There is an association between damage to neural progenitor cells (NPC) and neurocognitive dysfunction. NPC are similarly known to play an important role in recovery from damage to the brain, including radiation-induced damage. However NPC are extremely sensitive to radiation. In spite of this information, current RT planning techniques do not limit the radiation dose to the NPC containing regions. Recent human studies have demonstrated that it is possible to use intensity modulated radiation therapy to reduce the radiation dose to NPC containing regions during RT for brain tumors, without compromising coverage of the tumor. We hypothesize that NPC-sparing RT will reduce neurocognitive decline following treatment for brain tumors, without compromising tumor local control. However, there is conflicting data regarding the role of NPC in the development of glioblastoma multiforme (GBM). Some studies suggest that GBM are derived from NPC whereas others have associated NPC with improved tumor control following therapy for GBM. Prior to evaluation of neurocognitive outcomes with NPC-sparing RT, it is therefore imperative to evaluate whether NPC-sparing RT techniques lead to increased LR in the spared NPC containing niches of the brain.

The proposed study is designed to evaluate LR in the spared regions of the brain following NPC sparing RT in patients with newly diagnosed GBM. Our research will consist of 3 specific aims: 1) Determine the LR rate at 1 year in the spared NPC containing niches in patients treated with NPC sparing RT for GBM; 2) Quantify the extent of radiation dose sparing to the NPC containing regions that is possible without compromising tumor coverage in patients with GBM; 3) Determine if it is feasible to evaluate cognitive function prospectively in patients undergoing NPC sparing RT for GBM.

The long term goal of this research is to establish whether NPC sparing RT techniques improve neurocognitive outcomes compared to conventional RT for brain tumors. If the proposed study demonstrates that NPC sparing RT is not associated with increased LR in the spared regions of the brain compared to conventional RT, it will ideally serve as the foundation for a future multi-institutional randomized controlled trial comparing neurocognitive outcomes in patients treated with NPC-sparing RT versus conventional radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have newly diagnosed Glioblastoma Multiforme (GBM).
* Patient must have undergone surgical resection and must begin radiation within 12 weeks of this procedure.
* Patients must not have received previous irradiation to the brain.
* Patient must be at least 18 years of age
* Karnofsky performance status of greater than 60%
* Patient must receive temozolomide concurrent with and following radiation.
* If a woman is of child-bearing potential, a negative urine or serum pregnancy test must be demonstrated prior to treatment. Women of childbearing potential and men must agree to use adequate contraception for the duration of study participation and for up to 12 weeks following the study. Should a women become pregnant or suspect she is pregnant while participating in this study she should inform her treating physician immediately.
* Patient must have the ability to understand and the willingness to sign a written informed consent document.
* All patients must be informed of the investigational nature of this study and must be given written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients may not be receiving any other agents to treat their GBM
* No prior malignancy except for adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, or other cancer from which the patient has been disease free for at least 2 years.
* Patients with any other uncontrolled illness will be excluded.
* Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and up to 12 weeks after the study are excluded. This applies to any woman who has not experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months). Male subjects must also agree to use effective contraception for the same period as above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-12-27 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Redmond, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were screen failures
Groups:
- Neural Progeniter Cell Sparing Radiation With Temozolomide: All subjects are treated with neural progenitor cell sparing radiation to 60 Gy in 2 Gy per day, 30 fractions Concurrent and adjuvant temozolomide chemotherapy
  Radiation: Patients will be treated to a total dose of 60 Gy with a once daily fractionation schedule of 2 Gy per fraction, administered five days per week. All patients will undergo CT simulation with intravenous contrast. In addition they will undergo MRI simulation with both T1 with gadolinium as well as FLAIR sequences. They will be treated in a supine position using an aquaplast mask system for immobilization. CT image data will be reconstructed in approximately 3 mm slice thickness and manually coregistered with T1 post-gadolinium and FLAIR sequence MRI.
  Chemotherapy: Temozolomide
Period: Overall Study
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 58 [35 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Education [Median (Full Range); unit: years] — Number of years of education
  years | 16 [8 to 22]
Education [Count of Participants; unit: Participants] — Number of participants with greater than 12 years of education
  Participants | 20
Mini-Mental State Exam (MMSE) [Median (Full Range); unit: score on a scale] — The MMSE is a questionnaire used to measure cognitive impairment. The score ranges from 0-30 with a higher score, reflecting less impairment. Degree of impairment is interpreted by the following scores: 25-30= Questionably significant, 20-25= mild, 10-20= moderate, 0-10= severe.
  score on a scale | 26 [0 to 30]
Multifocal Tumor [Count of Participants; unit: Participants] | 6
MGMT promoter methylation [Count of Participants; unit: Participants]
  Positive | 8
  Negative | 14
  Unknown | 8
Resection extent [Count of Participants; unit: Participants]
  Gross total resection | 17
  Subtotal resection | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Recurrence in the Spared NPC Niches
Description: Number of participants with local recurrence (LR) at 1 year in the spared neural progenitor cell (NPC) containing niches of the brain in patients treated with NPC sparing radiation therapy (RT) plus temozolomide for newly diagnosed glioblastoma multiforme (GBM). Local recurrence in spared area is defined as development of a new regions of T1 post gadolinium enhancement.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 30
Participants | 0

2. Secondary Outcome: Extent of NPC Sparing
Description: The extent of NPC-sparing will be recorded for each patient. Patients will be binned into 4 groups according to the volume of NPC region that receives a certain dose as follows: 1) V5Gy≤50%; 2) V5Gy ≤20%; 3) V10Gy≤20%; 4) Doses higher than levels 1-3.
Time Frame: 1 year
Population: Data was not collected for this outcome measure
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 0

3. Secondary Outcome: Distance of Tumor to Spared NPC Niches
Description: The X-, Y-, and Z- coordinate distances in centimeters will be recorded from the most proximal point of the planning tumor volume to the closest point of the spared NPC-containing niche.
Time Frame: 1 year
Population: Data was not collected for this outcome measure.
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Neurocognitive Function as Measured by Wechsler Adult Intelligence Scale Fourth Edition (WAIS-IV) Coding Subtest
Description: Change in mean score of neurocognitive function (processing speed) as measured by WAIS-IV (Coding subtest) in patients treated with NPC sparing radiation for newly diagnosed GBM. The coding subtest of WAIS-IV is a visual, paper and pencil task that requires individuals to match numbers with symbols based on a "key" at the top of the page (Coding) by drawing the correct symbol in the boxes provided. Coding measures visual processing speed, short-term visual memory, and the ability to shift the eyes efficiently back and forth between the "key" and the responses. This task requires fine motor skills (using a pencil) but does not require expressive language. Minimal demands are placed on receptive language. This task also assesses the ability to sustain focus and effort for a two minutes. The score is the total number of correct responses within a given time frame, which ranges from 0-135. A higher score reflects a better outcome. A negative value for change reflects a worse outcome.
Time Frame: Change from baseline to 6 months
Population: Paired baseline and follow-up scores were only available in 14/30 participants.
Measure: Mean (95% Confidence Interval); unit: correct responses
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 14
correct responses | -6.9 [-12.9 to -0.8]

5. Secondary Outcome: Change in Neurocognitive Function as Measured by Trail Making Test
Description: Change in mean score of neurocognitive function as measured by Trail Making test Parts A and B in patients treated with NPC sparing radiation for newly diagnosed GBM. The Trail making score is the number of seconds spent connecting numbered circles (1-13) to circles containing letters of the alphabet (A-L) in alternating sequential order. Score ranges from 0-150 for Part A and 0-300 for Part B. A higher score reflects greater neurocognitive impairment. Therefore, a negative value for change reflects an improvement in this measure, whereas a positive value reflects worsening impairment.
Time Frame: Change from baseline to 6 months
Population: Paired baseline and follow-up scores were only available in 12/30 participants.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 12
seconds
  Trail Making Test Part A | 20.6 [-21.4 to 62.6]
  Trail Making Test Part B | -14.7 [-59.8 to 30.5]

6. Secondary Outcome: Change in Neurocognitive Function (Verbal Fluency) as Measured by Controlled Oral Word Association Test (COWAT)
Description: Change in neurocognitive function (verbal fluency) as measured by COWAT in patients treated with NPC sparing radiation for newly diagnosed GBM. COWAT assesses verbal fluency by asking the participant to produce words for three designated letters. The test score is the total number of different words produced for all three letters. A higher score reflects a better outcome. Therefore, a positive value for change reflects an improvement in this measure.
Time Frame: Change from baseline to 6 months
Population: Paired baseline and follow-up scores were only available in 14/30 participants.
Measure: Mean (95% Confidence Interval); unit: words
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 14
words | 2.6 [-2.8 to 8.1]

7. Secondary Outcome: Change in Neurocognitive Function (Total Recall, Delayed Recall, Recognition Discrimination) as Measured by Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: Change in total recall, delayed recall, and recognition discrimination index as measured by HVLT-R in patients treated with NPC sparing radiation for newly diagnosed GBM. 12-item word list, composed of four words from each of the three semantic categories which the patient must learn over three trials. For each trial, the subject is instructed to listen carefully as the examiner reads the word list and attempt to memorize the words. The score for total recall is the sum of all the correctly-recalled words from each trial, for a maximum of 36. Delayed recall is assessed as the number of words freely recalled 20-25 minutes after the learning trials. Recognition is assessed after 20-25 minutes where the patient is read 24 words and is asked to say "yes" after words from the recall list (12 targets) and "no" after other words (12 distractors). RDI is the number of recalled target words minus the number of recalled distractor words. A higher score reflects a better outcome.
Time Frame: Change from baseline to 6 months
Population: Paired baseline and follow-up scores were only available in 14/30 participants.
Measure: Mean (95% Confidence Interval); unit: words
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 14
words
  Total recall | -1.4 [-4.1 to 1.3]
  Delayed recall | -0.6 [-2.4 to 1.1]
  Recognition Discrimination Index (RDI) | -0.3 [-1.4 to 0.8]

8. Secondary Outcome: Radiation Dose to Spared NPC Region
Description: The mean radiation dose (cGy) to spared NPC region (hippocampus, subventricular zone [SVZ]) in reference to site of lesion.
Time Frame: Day 1 of radiation therapy
Measure: Mean (Full Range); unit: centigray (cGy)
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 30
centigray (cGy)
  Hippocampus (Ipsilateral) | 4906 [90 to 6139]
  Hippocampus (Contralateral) | 1652 [87 to 3584]
  Hippocampus (Bilateral) | 3473 [88 to 4820]
  SVZ (Ipsilateral) | 4181 [605 to 5970]
  SVZ (Contralateral) | 1986 [440 to 5358]
  SVZ (Bilateral) | 3096 [601 to 5481]

9. Secondary Outcome: Volume (cc) of "NPC for Sparing" Region
Description: The volume of the "NPC_for_sparing" region as collected using the Pinnacle treatment planning system.
Time Frame: day 1 of radiation therapy
Population: Data was not collected for this outcome measure
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 years (median follow-up time was 15.8 months)
Arm/Group | Neural Progeniter Cell Sparing Radiation With Temozolomide
All-Cause Mortality (participants affected / at risk) | 27/30
Serious Adverse Events (participants affected / at risk) | 17/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neural Progeniter Cell Sparing Radiation With Temozolomide (N=30)
Hospital admission for anticoagulation of venous thrombosis due to disease progression (Nervous system disorders) | 4 (4)
Hospital admission for craniotomy for removal of tumor from disease progression. (Nervous system disorders) | 1 (1)
Death due to disease progression. (Nervous system disorders) | 5 (5)
Hospital admission for pneumonia. (Infections and infestations) | 1 (1)
ER treatment for multifocal hemmorrhage due to head injury from fall. (Injury, poisoning and procedural complications) | 1 (1)
Hospital admission for progressive confusion. Treated for pneumatosis. (Infections and infestations) | 1 (1)
Patient report of melanoma. Subsequently diagnosed mild/moderate melanocytic dysplasia. (Skin and subcutaneous tissue disorders) | 1 (1)
ER due to seizure ending in car accident (Nervous system disorders) | 1 (1)
Admission to surgery of tumor within treatment field for glioblastoma. (Nervous system disorders) | 1 (1)
ER due to disorientation thought to be minor seizure. (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neural Progeniter Cell Sparing Radiation With Temozolomide (N=30)
Fatigue (General disorders) | 20
diarrhea (Gastrointestinal disorders) | 13
aphasia (Nervous system disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT01478854/Prot_SAP_000.pdf